CLINICAL TRIAL: NCT01635114
Title: Evaluate the Effects of resVidaTM on Liver Fat Content, Body Fat Distribution and Insulin Sensitivity
Brief Title: Effect of resVida on Liver Fat Content
Acronym: resVida NAFL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Norbert Stefan, Professor Dr. med., University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-12-10-RESV
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Elevated Liver Fat Content and Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- resVida (resveratrol) (Active Comparator)
  Interventions: Dietary Supplement: resveratrol
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: resveratrol — 150 mg resVida per day for 12 weeks
  Arms: resVida (resveratrol)
Dietary Supplement: Placebo — Placebo for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of the antioxidant "resveratrol" on liver fat content, body-composition and insulin sensitivity

Resveratrol is found in grape skin, wine, peanuts, and mulberries and is thought to have health benefits such as improving fat metabolism, insulin action, and possibly extending lifespan. resVida™ is the name for the dietary supplement containing the natural antioxidant "resveratrol". resVida™ will be supplied by DSM Nutritional Products, Ltd.

resVida™ is considered a dietary supplement, and therefore it is not an approved drug by German Authority. It is regulated like a food. The makers of resVida™ make no claim that this supplement is meant to treat any ailment.

This study is designed to investigate the health benefits of resveratrol.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male and female
* Age: 18 years - 70 years (inclusive)
* Overweight and obese (BMI ≥>27 mg/kg2)
* HOMA-IR ≥>2.0
* Negative urine pregnancy test
* Acceptable to be taking the oral contraceptive pill or other methods of birth control (surgical sterility, double barrier methods, intrauterine contraceptive device, lifestyle with a personal choice of abstinence, vasectomy of sexual partner at least 3 months prior to enrolment in combination with barrier methods)
* Willingness and ability to give written informed consent and willingness and ability to understand, to participate and to comply with the study requirements.

Exclusion Criteria:

* Subjects who have liver cirrhosis
* Subjects with a further liver disease diagnosis (e.g. known M. Wilson, autoimmune hepatitis, primary sclerosing cholangitis)
* Subjects who were diagnosed with diabetes
* Current pregnancy or breast feeding (as determined by a pregnancy test); postmenopausal women taking oral hormone therapy.
* Delivery within the last year
* Changes in the dose or initiation of lipid altering medication within the preceding three months, such as statins, fibrates or systemic steroids
* Significant co-morbid inflammatory illnesses as as rheumatoid arthritis, chronic bowel disease, sarkoidosis etc.
* Contraindications to MR scanning - claustrophobia, cardiac pacemaker, ferromagnetic haemostatic clips in the central nervous system, metallic splinters in the eye, automatic cardioverter defibrillators, prosthetic heart valves, cochlear implants, insulin pumps and nerve stimulators, etc. or who do not fit into the MR machine due to severe adiposity
* Subjects with any medical condition that is judged by the investigators to be likely to interfere with the evaluation of the subject's safety and of the study outcome.
* Subjects with abnormalities in the safety profile judged by the investigators to be clinically significant.
* Subjects with ALT or AST > 2.5x of the upper reference limit (50 U/L respectively)
* Subjects on treatment with drugs that are strongly metabolized via CYP3A4 (e.g. alfentanil, astemizole, cisapride, cyclosporine, diergotamine, ergotamine, fentanyl, irinotecan, pimozide, quinidine, sirolimus, tacrolimus, terfenadine) and CYP2C9 (e.g. Phenytoin and Warfarin)
* Smokers (> 10 cigarettes per day)
* Regular drinkers of more than15g /day (e.g wine (0,1 l), 1 beer (0,33 l)
* History of, or current evidence of, abuse of alcohol or any drug substance, licit or illicit.
* Intake of over-the-counter (OTC) medication or any dietary supplement (except occasional paracetamol/aspirin, and multivitamin supplements) for the duration of the study.
* Poor compliers or subjects unlikely to attend.
* Receipt of any investigational products (e.g., drugs, supplements, dietary interventions) as part of a research study within 30 days of initial dose administration in this study.
* Blood donation (usually 550 ml) within the 12 week period before the initial study dose.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Liver fat content | 3 months
  Measured by 1H-MRS

SECONDARY OUTCOMES:
Body composition | 3 months
  Total body-, visceral- and abdominal subcutaneous fat mass and intramyocellular fat content by MR tomography and 1H-MRS
Insulin sensitivity | 3 months
  Fasting serum insulin - HOMA-IR Oral Glucose Tolerance Test (OGTT) Matsuda insulin sensitivity index)
Intima-media thickness | 3 months
  Of common carotid artery
Blood analytes | 3 months
  Blood biochemistry
Cardiorespiratory fitness | 3 months
  VO2max

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Stefan, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany